CLINICAL TRIAL: NCT05112120
Title: Exploiting Leading Edge 7T MRI Brain Imaging to Decipher Olumiant's Mode of Analgesic Action in Rheumatoid Arthritis
Acronym: SOAR
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: GN19RH319
Record Dates: First submitted 2021-10-01; First posted 2021-11-08 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained to allow analysis of inflmamatory markers considered importnat in Rheumatoid Arthritis.

GROUPS / COHORTS (1):
- Single centre single arm observational cohort: Olumiant (4mg) will be administered in line with standard of care guidance. This is the standard dose in line with license for use in active moderate to severe RA. A dose adjustment from 4mg to 2mg is permitted during the study depending on side-effects
  Interventions: Drug: Olumiant

INTERVENTIONS:
Drug: Olumiant — Olumiant (4mg) will be administered in line with standard of care guidance.
  Other Names: Baricitinib

SUMMARY:
The revolution in treatments for rheumatoid arthritis (RA) has transformed patient outcomes, but many patients continue to experience life disabling pain. Even those who achieve full disease remission with state-of-the-art treatments report substantially higher levels of pain when compared to the general population. Researchers believe this disconnect is due to the existence of pain sources that are in addition to those present in the joints. In particular, the central nervous system (CNS) may have an important role in determining RA pain.

According to a recent study, RA patients who received treatment with Olumiant (a Janus Kinase (JAK) inhibitor that works by interfering with the inflammatory processes that lead to the symptoms of RA) reported better and quicker pain improvements compared to those receiving other types of therapy. However, this could not be explained by levels of peripheral inflammation alone and remains to be fully understood. Investigators think this improvement may be related to the role of the JAK pathway in the brain and that inhibition of this pathway with Olumiant could normalise brain connectivity in respect to pain processing.

Advanced brain scanning methods have already helped to identify specific regions of the brain that are thought to be important in pain processing and peripheral inflammation; a) enhanced functional connectivity between the Default Mode Network (DMN) and insula and b) enhanced functional connectivity between the Dorsal Attention Network (DAN) and the left inferior parietal lobule (LIPL). This study aims to elucidate the mechanisms of analgesic action of Olumiant by examining changes in functional connectivity and glutamate levels within the CNS and exploring the relationship between MRI markers, pain, clinical phenotype and peripheral immune markers.

DETAILED DESCRIPTION:
Investigators believe that RA is a mixed pain state i.e. pain pathways exist in addition to established peripheral inflammatory nociceptive mechanisms. In particular, the central nervous system (CNS) may have an important role in determining RA pain. Recently this group were the first to delineate distinct neurobiological pain signatures in the brains of RA patients by employing 3T functional connectivity magnetic resonance imaging (fcMRI) - a recent adaptation of functional MRI data that examines the synchrony of neural activity which modulates the efficiency and extent of neuronal transmission between brain regions. Specifically, researchers identified and replicated two distinct pain signatures: a) enhanced functional connectivity between the Default Mode Network (DMN) and insula which was unrelated to levels of peripheral inflammation but, intriguingly, is an established neurobiological marker of fibromyalgia (an archetypal CNS determined chronic pain disorder) and b) enhanced functional connectivity between the Dorsal Attention Network (DAN) and the left inferior parietal lobule (LIPL)6 which was related to levels of peripheral inflammation.

Pre-clinical experiments have not only implicated the JAK- signal transducer and activator of transcription (STAT) pathway with peripheral immune system functioning but also the brain. In the CNS, this pathway promotes gene expression associated with inflammation which in turn generates pro-nociceptive cytokines such as TNFα. However, there is now also emerging evidence to support the pathway's direct role in synaptic transmission and neurotransmitter receptor modulation. Specifically, the JAK-STAT pathway appears important in N-methyl-d-aspartate (NMDA) related synaptic plasticity - a ubiquitous glutamate receptor of the human brain. Their induction is selectively blocked by JAK inhibitors and JAK2 knockdown abolishes NMDA functioning. Increases in glutamate and subsequent binding to NMDA receptors cause chaotic and incoherent neuronal functional activity. In human studies of fibromyalgia, we have consistently evidenced both elevated glutamate levels within the insula and dysfunctional neural connectivity. Moreover, this group have shown that fibromyalgia pharmacotherapy (pregablin), considered to reduce neural glutamate, rectifies both insular glutamate and pro-nociceptive brain functional connectivity (DMN-insula). JAK inhibition (JAKi) may facilitate the reduction of glutamate-NMDA binding and ultimately pain alleviation by normalising the functional activity of these same neural connections.

There are clear practical constraints of sampling fresh human brain tissue in order to interrogate these possible mechanisms. Instead, neurobiological surrogate imaging measures may be employed. Glasgow benefits from the only clinical based ultra-high resolution 7T MRI scanner in the UK. Unlike lesser resolutions, 7T can distinguish the resonance of glutamate from other metabolites and so more precisely quantify the chemical of interest. Further, the superior spatial resolution of 7T enhances capacity to indirectly measure neuronal functional connectivity.

Investigators hypothesise that Olumiant's mechanism of analgesic action is determined by at least two factors. The first is related to those pathways seen in fibromyalgia, mediated via DMN-insula connectivity and insular glutamate. The second is related to peripheral inflammation, mediated via DAN-LIPL.

The study objectives include: 1) To evaluate the effects of Olumiant on DMN-Insula connectivity and insular glutamate levels in RA (neurobiological markers of fibromyalgia). 2) To evaluate the effects of Olumiant on DAN-LIPL connectivity in RA (neurobiological marker of peripheral inflammation). 3) To explore the relationship between pain, clinical phenotype, peripheral immune markers and their change with MRI markers indicative of CNS pathway function. The study will involve participants aged over 18 years with RA who are scheduled to start outpatient Olumiant as part of standard clinical practice, and who meet the inclusion criteria and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years < 75 years.
* Clinical diagnosis of RA
* Selected to start Olumiant by their usual rheumatology clinical team in line with local guidance (previous failure of at least 2 DMARDs and moderate to severe disease active disease)
* Right-handed (to reduce neuroimaging heterogeneity)

Exclusion Criteria:

* Inability to provide written informed consent.
* Severe physical impairment (e.g. blindness, deafness, paraplegia).
* Pregnant or breast feeding.
* Contraindications to MRI (e.g. severe claustrophobia).
* Major confounding neurological disease including Multiple Sclerosis, Stroke, Traumatic Brain Injury, Parkinson's Disease, Alzheimer's Disease
* Previous targeted synthetic (e.g. Oluminant, tofacitinib) DMARD exposure.
* Co-morbid medical conditions that may significantly impair physical functional status
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., malignancy, psychosis, suicidal ideation)
* BMI > 40 or unable to lie comfortably in MRI

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active RA attending clinics in NHS Greater Glasgow and Clyde who are scheduled to begin Olumiant as part of their standard NHS clinical care will be asked to contribute to this study by their point of care team.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of Olumiant on DMN-Insula connectivity | 12 weeks
  To measure brain functional connectivity DMN- insula and DNA- LIPL as measured by 7T MRS
To evaluate the effects of Oluminant treatment on insular glutamate levels in RA (neurobiological markers of fibromyalgia). | 12 weeks
  To examine changes in the insular glutamate signal as measured by the 7T MRS

SECONDARY OUTCOMES:
Changes in clinical phenotype as measured by the EULAR Disease Activity Score (DAS28) | 12 weeks
  Changes in clinical phenotype as measured by the EULAR Disease Activity Score (DAS28) from week 0 to week 12
Changes in clinical phenotype as measured by the CDAI | 12 weeks
  Changes in clinical phenotype as measured by the Clinical Disease Activity Index from week 0 to week 12
Changes in clinical phenotype as measured by the SDAI | 12 weeks
  Changes in clinical phenotype as measured by the Simple Disease Activity Index from week 0 to week 12
Changes in sickness behaviour as measured by the 7-Day Symptom Diary (Number Rating Scale) | 12 weeks
  Changes in sickness behaviours as measured by the 7-Day Symptom Diary (Number Rating Scale) from week 0 to week 12
Changes in sickness behaviour as measured by the American College of Rheumatology Fibromyalgia Scale | 12 weeks
  Changes in fibromyalgia as measured by the American College of Rheumatology Fibromyalgia Scale from week 0 to week 12
Changes in sickness behaviour as measured by the McGill Pain Questionnaire | 12 weeks
  Changes in pain as measured by the McGill Pain Questionnaire from week 0 to week 12
Changes in sickness behaviour as measured by the Michigan Body Map Regional Pain | 12 weeks
  Changes in pain as measured by the Michigan Body Map Regional Pain from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Depression | 12 weeks
  Changes in depression as measured by the PROMIS-Depression from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Anxiety | 12 weeks
  Changes in anxiety as measured by the PROMIS-Anxiety from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Fatigue | 12 weeks
  Changes in fatigue as measured by the PROMIS-Fatigue from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Sleep related impairment | 12 weeks
  Changes in sleep as measured by the PROMIS-Sleep related impairment from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Physical functioning short form | 12 weeks
  Changes in physical functioning as measured by the PROMIS-Physical functioning short form from week 0 to week 12
Changes in sickness behaviour as measured by the PROMIS-Pain inference | 12 weeks
  Changes in pain interference as measured by the PROMIS-Pain inference from week 0 to week 12
Changes in sickness behaviour as measured by the Cognitive Failures Questionnaire | 12 weeks
  Changes in cognitive function as measured by the Cognitive Failures Questionnaire from week 0 to week 12
Changes in sickness behaviour as measured by the Sickness Questionnaire | 12 weeks
  Changes in sickness behaviours as measured by the Sickness Questionnaire from week 0 to week 12
Changes in joint inflammation as measured by the Synovitis score | 12 weeks
  Changes in joint inflammation as measured by the Synovitis score (from joint ultrasound) from week 0 to week 12
Changes in pain as measured by the Pain sensitivity variables | 12 weeks
  Changes in pain as measured by the Pain sensitivity variables (from Quantitative Sensory Testing measures) from week 0 to week 12
Changes in inflammation as measured by the Changes in inflammatory cytokines/chemokines | 12 weeks
  Changes in peripheral inflammation as measured by the changes in inflammatory cytokines/chemokines from week 0 to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Neil Basu, M.D Ph.D, Principal Investigator — University of Glasgow
Locations (1):
- NHS GG&C, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT05112120/Prot_SAP_001.pdf